CLINICAL TRIAL: NCT02519868
Title: Chemical Block and Electrical Stimulation of the Carotid Body to Treat Refractory Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER 227-15
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Neuromodulation; Local anaesthetics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental): Patients will have both interventions: electrical stimulation followed by chemical stimulation
  Interventions: Device: Electrical block; Device: Chemical block

INTERVENTIONS:
Device: Electrical block — Nerve stimulator switched on at an intensity of 5 mA for 15 minutes, with the needle tip positioned close to the carotid bifurcation with the aid of the echography
Device: Chemical block — Injection of lidocaine 1%, 15 mLs, with the needle tip positioned close to the carotid bifurcation, with the aid of the echography

SUMMARY:
High blood pressure, also referred to as hypertension, affects about 65 million people in the United States alone. Approximately 25 percent of people with hypertension cannot control their high blood pressure, despite the use of multiple medications. Recently, new evidence has demonstrated that the carotid body (CB) plays a role in essential refractory hypertension, possibly due to a deregulated, enhanced activity of this organ. Animal studies showed that CB de-afferentiation, through carotid sinus nerve denervation, leads to a long-term stable drop in blood pressure in spontaneously hypertensive rats. De-afferentiation may be performed either by injecting local anesthetics or by electrical stimulation. Both techniques are daily used in the operating theater to anesthetize nerves for a wide range of surgical procedures. We hypothesize that blocking CB with local anesthetics will result in a drop of the blood pressure in refractory hypertensive patients. We also want to test the idea that stimulating the CB with an electrical current will mislead the CB and will also result in a drop of the blood pressure.

DETAILED DESCRIPTION:
High blood pressure, also referred to as hypertension, affects about 65 million people in the United States alone. Approximately 25 percent of people with hypertension cannot control their high blood pressure, despite the use of multiple medications.

Recently, new evidence has demonstrated that the carotid body (CB) plays a role in essential refractory hypertension, possibly due to a deregulated, enhanced activity of this organ. Animal studies showed that CB de-afferentiation, through carotid sinus nerve denervation, leads to a long-term stable drop in blood pressure in spontaneously hypertensive rats. It has been further shown that hypertonicity of the CB leads to a sympathetic hyper-excitation in SH rats and causes an increased vasomotor tone, which in turn contributes to hypertension.

The increased knowledge about the role of the CB in essential hypertension has lead to the development of an implantable (via open surgery) pulse generator, which lead to significant decrease in blood pressure at 12 months. One-year results from 13 patients showed a 39 mmHg average decrease in systolic blood pressure and a 26 mmHg average decrease in diastolic blood pressure in early reports. Beside, the procedure is invasive and requires surgery under general anesthesia.

De-afferentiation may be performed either by injecting local anesthetics or by electrical stimulation. Both techniques are daily used in the operating theater to anesthetize nerves for a wide range of surgical procedures.

We hypothesize that blocking CB with local anesthetics will result in a drop of the blood pressure in refractory hypertensive patients. We also want to test the idea that stimulating the CB with an electrical current will mislead the CB and will also result in a drop of the blood pressure. Preliminary results will shed some light on the mechanism of action of the CB in refractory hypertension and will open the way to new therapeutical approaches such as development of new implantable devices through a transcutaneous approach.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age, inclusive;
* blood pressure not controlled despite 3 different anti-hypertensive drugs;
* minimal body weight of 70 kg.

Exclusion Criteria:

* history of neck surgery or radiotherapy;
* secondary hypertension;
* contraindications to regional anesthesia (e.g., allergy to local anesthetics, coagulopathy, bleeding diathesis, malignancy or infection in the area);
* pregnancy;
* severe respiratory disease;
* inability to understand the informed consent and demands of the study;
* patient refusal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 15 minutes after electrical block and 15 minutes after chemical block

SECONDARY OUTCOMES:
Heart rate | 15 minutes after each intervention
Presence of paraesthesia | During the procedure
Presence of dyspnea | During the procedure
Presence of Claude-Bernard-Horner Syndrome | During the procedure
Presence of hoarseness | During the procedure
Presence of hematoma | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, PD Dr, Principal Investigator — CHUV
Locations (1):
- Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] McBryde FD, Abdala AP, Hendy EB, Pijacka W, Marvar P, Moraes DJ, Sobotka PA, Paton JF. The carotid body as a putative therapeutic target for the treatment of neurogenic hypertension. Nat Commun. 2013;4:2395. doi: 10.1038/ncomms3395. PMID 24002774
- [Background] Alnima T, Scheffers I, De Leeuw PW, Winkens B, Jongen-Vancraybex H, Tordoir JH, Schmidli J, Mohaupt MG, Allemann Y, Kroon AA. Sustained acute voltage-dependent blood pressure decrease with prolonged carotid baroreflex activation in therapy-resistant hypertension. J Hypertens. 2012 Aug;30(8):1665-70. doi: 10.1097/HJH.0b013e3283551f10. PMID 22728906